CLINICAL TRIAL: NCT00171470
Title: The Role of Tegaserod Therapy in the Management of Dyspeptic Symptoms in Female Patients on Proton Pump Inhibitors for the Treatment of Heartburn.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHTF919DUS46
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-02-01 (Estimated); Status verified 2008-01

CONDITIONS: Dyspepsia
Keywords: dyspepsia; hearburn; female; PPI
MeSH Terms: conditions — Dyspepsia | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
Study to provide initial data to assess the safety and efficacy of tegaserod use in patients with dyspepsia that are being treated with proton pump inhibitors (PPI's) for heartburn.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years or older.
* Self-reported presence of symptoms consistent with dyspepsia (including mid-upper abdominal discomfort characterized by post prandial fullness, early satiety and bloating)
* Stable dose PPI therapy of at least 4 weeks

Exclusion Criteria:

* History of intestinal obstruction, symptomatic gallbladder disease, suspected sphincter of Oddi dysfunction, or of abdominal adhesions.
* Evidence that the dyspeptic symptoms are relieved by defecation and/or associated with a change in frequency or stool form.
* With a current most bothersome symptom of heartburn.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-04; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To determine whether tegaserod administered over 6 weeks results in improved dyspeptic symptoms characterized by epigastric discomfort vs placebo on patients taking PPIs for the treatment of heartburn (weekly global assessment)

SECONDARY OUTCOMES:
Comparison of tegaserod vs. placebo for individual symptoms severity scores of postmeal fullness, early fullness while eating, bloating, abdominal pain, nausea, vomiting, heartburn, regurgitation and constipation (daily assessment)
Quality of Life (weekly assessment)
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- http://www.novartisclinicaltrials.com/etrials/DiseaseID21/Dyspepsia-clinical-trials.go, East Hanover, New Jersey, United States

REFERENCES:
- See also: Novartis patient recruitment website — http://www.novartisclinicaltrials.com/etrials/DiseaseID21/Dyspepsia-clinical-trials.go